CLINICAL TRIAL: NCT03473353
Title: Doctor-Parent Interactions With Medical Scribes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin H. Levi, Professor, Departments of Humanities & Pediatrics, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00007664
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Burnout, Professional
Keywords: Medical Scribe; Outpatient; EHR
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric Clinicians (Other): Survey data will be gathered from pediatric clinicians and also parents of pediatric patients at two time periods. At baseline, no Medical Scribes will be working with the clinicians, and then several months later, data will be gathered when Medical scribes ARE working with clinicians.
  Interventions: Other: Medical Scribe

INTERVENTIONS:
Other: Medical Scribe — Trained Medical Scribes will be present in the exam room to take notes on the the electronic medical record so that clinicians can focus all their attention to the interaction with the patient and parent.

SUMMARY:
The purpose of the study is to collect outcomes related to a quality improvement project assessing the feasibility and effectiveness of a medical scribe program in which medical scribes accompany clinicians during their visits with patients. The medical scribes involved in the project are professional scribes and medical students who will accompany clinicians during patient visits and takes notes, enabling the clinician to engage more directly with the patient.

DETAILED DESCRIPTION:
The study has several specific objectives. This study aims to examine the impact of using medical scribes on (1) patient experience (e.g. patient satisfaction) (2) clinician experience (e.g. stress load, burnout, evaluation of the visit, amount of time spent after hours inputting notes), and (3) clinician-patient interaction (e.g. patient and clinician engagement during the visit).

ELIGIBILITY:
Provider Participants

Inclusion Criteria:

1. Attending clinicians with privileges at Penn State Hershey Children's Hospital and/or the Penn State Hershey Internal Medicine. This may include attending MDs or DOs and Nurse Practitioners (NPs).
2. Voluntary participation in the medical scribe QI project.
3. Consents to participate in the study.

Exclusion Criteria:

1. Clinician is not participating in the scribe project.
2. Clinician does not consent to participate in the research portion of this project.

Patient Participants

Inclusion Criteria:

1. Patient (if 18 years or older) or parent/guardian (P/G) of patient being seen by a participating clinician.
2. Patient was not seen by a resident or medical student prior to meeting with clinician.
3. English speaking/reading.
4. Patient or P/G has capacity to consent.

Exclusion Criteria:

1. Patient is seeing a clinician who has not consented to participate in the research portion of the study.
2. Non-English speaking/reading.
3. Patient or P/G lacks capacity to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 732 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Clinician Burnout | 1 year
  Survey questions will assess clinician burnout using validated measures.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Levi, M.D., Ph.D., Principal Investigator — Departments of Humanities & Pediatrics
Locations (1):
- Hope Drive Pediatric Clinic, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The study PI will share our study protocol, instruments, and published papers (which include our analytic approach).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study information will be shared upon request to the study PI (Levi), and will be available through 6-30-26.
Access Criteria: Any interested researcher should contact the PI at: BHLevi@psu.edu.

REFERENCES:
- See also: Manuscript on impact of scribe intervention on documentation — https://doi.org/10.1016/j.acap.2021.05.004
- See also: Manuscript on impact of scribe intervention on relative value units (RVUs) — https://doi.org/10.1016/j.acap.2020.05.009